CLINICAL TRIAL: NCT05486052
Title: Evaluation of the Effectiveness of Biofeedback Rehabilitation in Patients With Neurological Diseases
Brief Title: Rehabilitation With Biofeedback in Neurology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Justyna Leszczak, Principal Investigator, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: neurological rehabilitation
Record Dates: First submitted 2022-07-18; First posted 2022-08-03 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Rehabilitation; Biofeedback; Neurological Diseases
Keywords: Rehabilitation; Health-resort based rehabilitation; Conventional (traditional) rehabilitation; Lipid profile; Optical oximetry

STUDY DESIGN:
Intervention Model Description: Prior to the study, an assessment of the reliability, reproducibility and validity of the instrument will be conducted among healthy individuals followed by random selection into two groups (study group and control group)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Evaluation of reliability, repeatability and validity of devices among healthy subjects (Other): Evaluation of the reliability, repeatability and credibility of biofeedback-based devices such as Biometrics, Luna EMG, Vectis, Rotor and nIRS among healthy individuals
  Interventions: Other: Evaluation of reliability, repeatability and validity of devices among healthy subjects
- Biofeedback method and Health-resort based rehabilitation (Other): Health-resort based treatments supplemented with biofeedback training
  Interventions: Other: Biofeedback method and Health-resort based rehabilitation Health-resort based treatments supplemented with biofeedback training; Other: Health-resort based rehabilitation Control group - health-resort based treatments, without biofeedback training.
- Health-resort based rehabilitation (Other): Control group - health-resort based treatments, without biofeedback training.
  Interventions: Other: Health-resort based rehabilitation Control group - health-resort based treatments, without biofeedback training.

INTERVENTIONS:
Other: Evaluation of reliability, repeatability and validity of devices among healthy subjects — Evaluation of reliability, reproducibility and validity of devices among healthy subjects Prior to the study among individuals with neurological disorders, an evaluation of the reliability, repeatability and credibility of the devices to be included in the biofeedback rehabilitation and optical oximetry measurements will be carried out.
  The evaluation of the devices will be carried out by two independent researchers twice
  Arms: Evaluation of reliability, repeatability and validity of devices among healthy subjects
Other: Biofeedback method and Health-resort based rehabilitation Health-resort based treatments supplemented with biofeedback training — The rehabilitation programme will run for 3 weeks from Monday to Friday. Patients will receive: group and individual exercises (active and assisted exercises, manipulative exercises, PNF-based exercises, balance and breathing exercises), manual massages, physical treatments such as laser, whirlpool, mud packs, carbonic acid therapy , TENS therapy, BIO-V lamp, local cryotherapy.
  Health-resort based rehabilitation The rehabilitation programme will last 3 weeks from Monday to Friday. Patients will receive: group and individual exercises (active and assisted exercises, manipulative exercises, PNF-based exercises, balance and breathing exercises), manual massage, physical treatments such as laser, whirlpool, peat wraps, carbonic acid therapy , TENS therapy, BIO-V lamp, local cryotherapy.
  Arms: Biofeedback method and Health-resort based rehabilitation
Other: Health-resort based rehabilitation Control group - health-resort based treatments, without biofeedback training. — Health-resort based rehabilitation The rehabilitation programme will last 3 weeks from Monday to Friday. Patients will receive: group and individual exercises (active and assisted exercises, manipulative exercises, PNF-based exercises, balance and breathing exercises), manual massage, physical treatments such as laser, whirlpool, mud packs, carbonic acid therapy , TENS therapy, BIO-V lamp, local cryotherapy
  Arms: Biofeedback method and Health-resort based rehabilitation; Health-resort based rehabilitation

SUMMARY:
The research will aim to evaluate biofeedback rehabilitation and optical oximetry assessment in neurological patients and the influence of blood parameters on the effect of the rehabilitation carried out.

An additional aim will be to evaluate components of body weight, lifestyle, dietary habits, assessment of mental state, quality of life among the study subjects.

DETAILED DESCRIPTION:
Prior to the study, an assessment of the reliability, reproducibility and validity of the devices among healthy individuals will be carried out.

The subjects will be allocated, by random selection, to two groups:

- a study group (60 subjects) - following a conventional rehabilitation programme supplemented additionally with biofeedback training

Study subjects:

* Post-stroke condition;
* Craniocerebral trauma;
* Multiple Sclerosis;
* Cerebral Palsy;
* Parkinson's disease
* Complete or partial spinal cord injury The group of subjects are patients staying at the Health Resort and Rehabilitation Hospital in Iwonicz Zdrój. The subjects will have a comprehensive rehabilitation with additional exercises/therapies using modern equipment (Biometrics, Luna EMG, HEG, Vectis, Rotor) with the biofeedback method (the study group). Control group - standard sanatorium rehabilitation programme without biofeedback exercises. Patients will have an ongoing rehabilitation period in hospital (3 weeks). The first examination will be carried out on the day of admission to hospital, the second examination on the day of discharge and, 3 months after leaving hospital, the third examination (follow-up) during the follow-up visit.

In addition, subjects will have blood tests taken, such as blood count, GL, TG, TC, HDL, LDL, CRP, serum glucose, cytokines, myokines, markers found in neurological diseases, and optical oximetry (nIRS device) will be measured.

Measurements will be taken three times for all subjects:

* assessment of hand muscle strength
* ranges of motion of hand joints
* analysis of body composition using the Tanita 780 MA analyser (body fat, lean tissue, muscle tissue, body water content
* calculated body mass index (BMI)
* examination of deep sensation (mirror test)
* evaluation of the effects of rehabilitation
* functional capacity - Barthel index, ADL
* Ashworth muscle tension (spasticity)
* Manual dexterity of the hand using the Box and Blocks test
* grip function of the hand according to Franchay scale
* Motor abilities of the hand according to Fugl-Meyer Motor Assessment Scale for Upper Extremity

  * EDSS scale
  * WHOQOL-BREF quality of life scale
  * Berg scale
  * GMFCS scale
  * MACS scale
  * PEDI scale
  * GMFM scale
* Assessment of health related behaviours, eating habits, lifestyle, quality of life - standardised questionnaires. In addition, participants in the study will complete a survey questionnaire containing information on, among other things, education, marital status, place of residence.

ELIGIBILITY:
Inclusion Criteria:

* informed, voluntary consent of the patient
* age 21-75 years
* elementary (basic) gripping ability
* degree of paresis of the upper limb and hand 4 -5 on the Brunnström scale
* degree of disability on the Rankin scale 3
* spastic tension of the upper limb, paresis hand not more than 3 on the modified Ashworth scale - current health condition confirmed by a medical examination, allowing participation in tests and exercises

Test persons:

* after a stroke;
* Craniocerebral trauma;
* Multiple sclerosis;
* Cerebral Palsy;
* Parkinson's disease
* Total or partial spinal cord injury

Exclusion Criteria:

* lack of informed, voluntary consent of the patient

  * second or subsequent stroke, hemorrhagic stroke, stroke of the brainstem and cerebellum
  * disorders of higher mental functions limiting comprehension and carrying out tasks during exercises
  * visual field disturbances
  * mechanical and thermal injuries that may limit the grasping function of the hand
  * concomitant neurological, rheumatological and orthopedic diseases, including permanent contractures that may affect the grasping ability and locomotion
  * unstable medical condition
* metal implants, electronic implants, menstruation in women, epilepsy,
* failure to complete a 3-week rehabilitation stay

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
assessment of prioprioception (deep sensation) | research among healthy people, during studies from the 3rd to the 5th year of studies
  Measurement performed on the Luna EMG device, selected range of motion with eyes closed 60 degrees elbow joint flexion
assessment of prioprioception (deep sensation) | First examination - before the start of the rehabilitation program;
  Measurement performed on the Luna EMG device, selected range of motion with eyes closed 60 degrees elbow joint flexion
assessment of prioprioception (deep sensation) | Second examination - at the end of the three-week program
  Measurement performed on the Luna EMG device, selected range of motion with eyes closed 60 degrees elbow joint flexion
assessment of muscle tone (spasticity) | research among healthy people, during studies from the 3rd to the 5th year of studies
  measurement performed on the Luna EMG machine, range of motion from 0 to 90 degrees elbow joint flexion
assessment of muscle tone (spasticity) | First examination - before the start of the rehabilitation program;
  measurement performed on the Luna EMG machine, range of motion from 0 to 90 degrees elbow joint flexion
assessment of muscle tone (spasticity) | Second examination - at the end of the three-week program
  measurement performed on the Luna EMG machine, range of motion from 0 to 90 degrees elbow joint flexion
ranges of movements in the shoulder joint | research among healthy people, during studies from the 3rd to the 5th year of studies
  measurements performed on the Vectis , shoulder joint range of motion: flexion to 170, extension to 170
ranges of movements in the shoulder joint | First examination - before the start of the rehabilitation program;
  measurements performed on the Vectis , shoulder joint range of motion: flexion to 170, extension to 170
ranges of movements in the shoulder joint | Second examination - at the end of the three-week program
  measurements performed on the Vectis , shoulder joint range of motion: flexion to 170, extension to 170
Hand grip strength | First examination - before the start of the rehabilitation program;
  measurements to be performed with a dynamometer The dynamometer registers strength lower than up to 90 kg,
Hand grip strength | Second examination - at the end of the three-week program
  measurements to be performed with a dynamometer The dynamometer registers strength lower than up to 90 kg,
pinching strength of the fingers | First examination - before the start of the rehabilitation program
  measurements to be performed with a pinch meter. The pinch meter registers strength lower than up to 22 kg.
pinching strength of the fingers | Second examination - at the end of the three-week program
  measurements to be performed with a pinch meter. The pinch meter registers strength lower than up to 22 kg.
Hand grip strength | research among healthy people, during studies from the 3rd to the 5th year of studies
  measurements to be performed with a dynamometer The dynamometer registers strength lower than up to 90 kg,
pinching strength of the fingers | research among healthy people, during studies from the 3rd to the 5th year of studies
  measurements to be performed with a pinch meter. The pinch meter registers strength lower than up to 22 kg.
optical oximetry | research among healthy people, during studies from the 3rd to the 5th year of studies
  measurement performed with nIRS device, ranges: near infrared light (700-1300 nm) for oxyhaemoglobin (O2Hb) and deoxyhaemoglobin (HHb)
optical oximetry | First examination - before the start of the rehabilitation program
  measurement performed with nIRS device, ranges: near infrared light (700-1300 nm) for oxyhaemoglobin (O2Hb) and deoxyhaemoglobin (HHb)
optical oximetry | Second examination - at the end of the three-week program
  measurement performed with nIRS device, ranges: near infrared light (700-1300 nm) for oxyhaemoglobin (O2Hb) and deoxyhaemoglobin (HHb)
Change Body composition assessment (fat mass, visceral fat level , muscle tissue, fat free mass , water content in the body) subjected to bioelectrical impedancy analysis - Tanita 780. | First examination - before the start of the rehabilitation program
  Assessment of body composition (bioelectrical impedancy analysis - Tanita 780) Change from Baseline body composition at 3 weeks between baseline, after the end of protocol treatment
Change Body composition assessment (fat mass, visceral fat level , muscle tissue, fat free mass , water content in the body) subjected to bioelectrical impedancy analysis - Tanita 780. | Second examination - at the end of the three-week program
  Assessment of body composition (bioelectrical impedancy analysis - Tanita 780)
Ranges of motion in the joints of the upper limb | research among healthy people, during studies from the 3rd to the 5th year of studies
  with the use of R 500 goniometer; the device operates with an accuracy up to one degree.
Ranges of motion in the joints of the upper limb | First examination - before the start of the rehabilitation program
  with the use of R 500 goniometer; the device operates with an accuracy up to one degree.
Ranges of motion in the joints of the upper limb | Second examination - at the end of the three-week program
  with the use of R 500 goniometer; the device operates with an accuracy up to one degree.
EMG of the extensors and flexors of the joints in the upper limb | research among healthy people, during studies from the 3rd to the 5th year of studies
  EMG of the extensors and flexors of the upper limb joints - Biometrics and Luna device
EMG of the extensors and flexors of the joints in the upper limb | First examination - before the start of the rehabilitation program
  EMG of the extensors and flexors of the upper limb joints - Biometrics and Luna device
EMG of the extensors and flexors of the joints in the upper limb | Second examination - at the end of the three-week program
  EMG of the extensors and flexors of the upper limb joints - Biometrics and Luna device

SECONDARY OUTCOMES:
Assessment of functional status was assessed using the Barthel Index. The subjects could score the maximum of 100 points. | First examination - before the start of the rehabilitation program
  Activities of daily living were assessed using Barthel Index. The subjects could score the maximum of 100 points.
  A maximum of 100 points can be obtained on the Barthel scale. There are three assessment ranges: getting from 0 to 20 points. means total dependence, from 20 to 80 points. means that to some extent the patient needs help from others, and the assessment in the border is 80 to 100 points. means that with a little help the patient can function alone.
  0-20 points patient's condition "light" 21-85 points - "medium-heavy" patient condition 86-100 points - patient condition "very heavy"
Assessment of functional status was assessed using the Barthel Index. The subjects could score the maximum of 100 points. | Second examination - at the end of the three-week program
  Activities of daily living were assessed using Barthel Index. The subjects could score the maximum of 100 points.
  A maximum of 100 points can be obtained on the Barthel scale. There are three assessment ranges: getting from 0 to 20 points. means total dependence, from 20 to 80 points. means that to some extent the patient needs help from others, and the assessment in the border is 80 to 100 points. means that with a little help the patient can function alone.
  0-20 points patient's condition "light" 21-85 points - "medium-heavy" patient condition 86-100 points - patient condition "very heavy"
Balance was assessed using Berg Balance Scale (BBS) | First examination - before the start of the rehabilitation program
  Balance was assessed using Berg balance scale (BBS)
  Berg Balance Scale
  Description:
  14-item scale designed to measure balance
  (1. Sitting to standing 2. Standing unsupported 3. Sitting unsupported 4. Standing to sitting 5. Transfers 6. Standing with eyes closed 7. Standing with feet together 8. Reaching forward with outstretched arm 9. Retrieving object from floor 10. Turning to look behind 11. Turning 360 degrees 12. Placing alternate foot on stool 13. Standing with one foot in front 14. Standing on one foot)
  Scoring: A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Score the LOWEST performance. Total Score = 56
  Interpretation: 41-56 = independent 21-40 = walking with assistance 0 -20 = wheelchair bound
Balance was assessed using Berg Balance Scale (BBS) | Second examination - at the end of the three-week program
  Balance was assessed using Berg balance scale (BBS)
  Berg Balance Scale
  Description:
  14-item scale designed to measure balance
  (1. Sitting to standing 2. Standing unsupported 3. Sitting unsupported 4. Standing to sitting 5. Transfers 6. Standing with eyes closed 7. Standing with feet together 8. Reaching forward with outstretched arm 9. Retrieving object from floor 10. Turning to look behind 11. Turning 360 degrees 12. Placing alternate foot on stool 13. Standing with one foot in front 14. Standing on one foot)
  Scoring: A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Score the LOWEST performance. Total Score = 56
  Interpretation: 41-56 = independent 21-40 = walking with assistance 0 -20 = wheelchair bound
Assessment of muscle tone (spasticity) was examined with modified Ashworth scale. | First examination - before the start of the rehabilitation program
  Increased muscle tone (spasticity) was examined with modified Ashworth scale. This is a six-point scale modified to include grade 1.
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Assessment of muscle tone (spasticity) was examined with modified Ashworth scale. | Second examination - at the end of the three-week program
  Increased muscle tone (spasticity) was examined with modified Ashworth scale. This is a six-point scale modified to include grade 1.
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Assessment of paretic limb function was assessed using the Brunnström scale. | First examination - before the start of the rehabilitation program
  Motor performance (function) of extremities was assessed using Brunnström scale. This is a six-point scale designed to assess performance (function) of paretic extremities
Assessment of paretic limb function was assessed using the Brunnström scale. | Second examination - at the end of the three-week program
  Motor performance (function) of extremities was assessed using Brunnström scale. This is a six-point scale designed to assess performance (function) of paretic extremities
Assessment of disability level, using the modified Rankin scale (MRS) | First examination - before the start of the rehabilitation program
  Assessment of disability using the modified Rankin scale (MRS)
  Score Description 0 - No symptoms at all
  1- No significant disability despite symptoms; able to carry out all usual duties and activities 2 - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance 3 - Moderate disability; requiring some help, but able to walk without assistance 4 - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance 5 - Severe disability; bedridden, incontinent and requiring constant nursing care and attention 6 - Dead TOTAL (0-6): _______
Assessment of disability level, using the modified Rankin scale (MRS) | Second examination - at the end of the three-week program
  Assessment of disability using the modified Rankin scale (MRS)
  Score Description 0 - No symptoms at all
  1- No significant disability despite symptoms; able to carry out all usual duties and activities 2 - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance 3 - Moderate disability; requiring some help, but able to walk without assistance 4 - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance 5 - Severe disability; bedridden, incontinent and requiring constant nursing care and attention 6 - Dead TOTAL (0-6): _______
Manual skills, assessed with Box and Blocks test; | First examination - before the start of the rehabilitation program
  The test uses a wooden box, divided into two equal parts by a partition, as well as 150 blocks. The subject moves as many blocks as possible from one part of the box to the other during 60 seconds.
Manual skills, assessed with Box and Blocks test; | Second examination - at the end of the three-week program
  The test uses a wooden box, divided into two equal parts by a partition, as well as 150 blocks. The subject moves as many blocks as possible from one part of the box to the other during 60 seconds.
Handgrip function, according Franchay scale | First examination - before the start of the rehabilitation program
  The scale consists of 7 tasks (pass/fail grading); the patient is awarded 1 point for each activity performed successfully, or 0 points for a failure to perform. The maximum score of seven points may be achieved for the performance of the tasks. Higher score corresponds to better manual skills. The scale measures the proximal control of the upper limb and the manual skills.
Handgrip function, according Franchay scale | Second examination - at the end of the three-week program
  The scale consists of 7 tasks (pass/fail grading); the patient is awarded 1 point for each activity performed successfully, or 0 points for a failure to perform. The maximum score of seven points may be achieved for the performance of the tasks. Higher score corresponds to better manual skills. The scale measures the proximal control of the upper limb and the manual skills.
Motor capacities of the upper limb, according to Fugl-Meyer Motor Assessment Scale | First examination - before the start of the rehabilitation program
  Fugl-Meyer Motor Assessment Scale for Upper Extremity is a comprehensive tool enabling measurement of motor function; it comprises 33 motor tasks, designed to assess general movements, precision movements, grip, coordination and speed. It is also possible to perform H subgroup tests - assessing superficial and deep sensibility, and J subgroup tests - for range of passive motion and pain induced by such movements.
  Individual tasks are assessed on a scale 0-2 0 - impossible task
  1. - task partially completed,
  2. - task completed correctly The higher the score, the better.
Motor capacities of the upper limb, according to Fugl-Meyer Motor Assessment Scale | Second examination - at the end of the three-week program
  Fugl-Meyer Motor Assessment Scale for Upper Extremity is a comprehensive tool enabling measurement of motor function; it comprises 33 motor tasks, designed to assess general movements, precision movements, grip, coordination and speed. It is also possible to perform H subgroup tests - assessing superficial and deep sensibility, and J subgroup tests - for range of passive motion and pain induced by such movements.
  Individual tasks are assessed on a scale 0-2 0 - impossible task
  1. - task partially completed,
  2. - task completed correctly The higher the score, the better.
Gross Motor Function Classification System (GMFCS) | First examination - before the start of the rehabilitation program
  the GMFCS is a 5-step assessment system for functioning and mobility in daily life.
Gross Motor Function Classification System (GMFCS) | Second examination - at the end of the three-week program
  the GMFCS is a 5-step assessment system for functioning and mobility in daily life.
Manual Ability Classification System (MACS) | First examination - before the start of the rehabilitation program
  The Manual Ability Classification System (MACS) describes how children with cerebral palsy use their hands when handling objects in everyday life. The MACS includes five levels. The assignment of a specific level to a child is based on the child's initiated activity during which they use objects, and whether the child needs the help of another person or the adaptation of equipment to be able to use them in everyday activities. The MACS booklet also describes the differences between adjacent levels to make it easier to determine which level best describes the child's ability to use objects.
Manual Ability Classification System (MACS) | Second examination - at the end of the three-week program
  The Manual Ability Classification System (MACS) describes how children with cerebral palsy use their hands when handling objects in everyday life. The MACS includes five levels. The assignment of a specific level to a child is based on the child's initiated activity during which they use objects, and whether the child needs the help of another person or the adaptation of equipment to be able to use them in everyday activities. The MACS booklet also describes the differences between adjacent levels to make it easier to determine which level best describes the child's ability to use objects.
Changes in blood parameter: HDL | First examination - before the start of the rehabilitation program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  HDL level:
  Men:
  Less than 35 mg / dL (0.9 mmol / L) high risk of heart disease.
  Women:
  Lower than 45 mg / dL (1.2 mmol / L) high risk of heart disease. 60 mg / dL (1.56 mmol / L) and above. High HDL cholesterol.
Changes in blood parameter: HDL | Second examination - at the end of the three-week program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  HDL level:
  Men:
  Less than 35 mg / dL (0.9 mmol / L) high risk of heart disease.
  Women:
  Lower than 45 mg / dL (1.2 mmol / L) high risk of heart disease. 60 mg / dL (1.56 mmol / L) and above. High HDL cholesterol.
Changes in blood parameter: LDL | First examination - before the start of the rehabilitation program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  LDL level:
  Less than 100 mg / dL (2.6 mmol / L) Norm 100 - 129 mg / dL (2.63.34 mmol / L) Above the norm 130 - 159 mg / dL (3.36 - 4.13 mmol / L) Limit 160 - 189 mg / dL (4.14 - 4.90 mmol / L) High 190 mg / dL (4.91 mmol / L) and above Very high
Changes in blood parameter: LDL | Second examination - at the end of the three-week program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  LDL level:
  Less than 100 mg / dL (2.6 mmol / L) Norm 100 - 129 mg / dL (2.63.34 mmol / L) Above the norm 130 - 159 mg / dL (3.36 - 4.13 mmol / L) Limit 160 - 189 mg / dL (4.14 - 4.90 mmol / L) High 190 mg / dL (4.91 mmol / L) and above Very high
Changes in blood parameter: total cholesterol | First examination - before the start of the rehabilitation program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  Total Cholesterol level:
  Less than 200 mg / dL (5.17 mmol / L) Norm 200 - 239 mg / dL (5.17 - 6.18 mmol / L) Elevated level 240 mg / dL (6.21 mmol / L) High risk of heart disease
Changes in blood parameter: total cholesterol | Second examination - at the end of the three-week program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  Total Cholesterol level:
  Less than 200 mg / dL (5.17 mmol / L) Norm 200 - 239 mg / dL (5.17 - 6.18 mmol / L) Elevated level 240 mg / dL (6.21 mmol / L) High risk of heart disease
Assessment of WHR | First examination - before the start of the rehabilitation program
  The type of obesity is assessed with the so-called waist-to-hip ratio (WHR), which shows the proportion of waist circumference and hip circumference. WHR specifies the location of excessive fat and makes it possible to identify two main types of obesity: visceral obesity (characteristic for men), connected with accumulation of fat in the abdominal cavity and upper part of the body, and gynoid obesity (gluteal-femoral), more common in women.
Assessment of WHR | Second examination - at the end of the three-week program
  The type of obesity is assessed with the so-called waist-to-hip ratio (WHR), which shows the proportion of waist circumference and hip circumference. WHR specifies the location of excessive fat and makes it possible to identify two main types of obesity: visceral obesity (characteristic for men), connected with accumulation of fat in the abdominal cavity and upper part of the body, and gynoid obesity (gluteal-femoral), more common in women.
Assessment of metabolic syndrome | First examination - before the start of the rehabilitation program
  Metabolic syndrome (polymetabolic syndrome, syndrome X, insulin resistance syndrome, Reaven syndrome) - a set of interrelated factors significantly increasing the risk of atherosclerosis and type 2 diabetes, as well as their vascular complications.
  Abdominal (central) obesity
  At least three of the following five abnormalities must be identified to formulate a diagnosis:
  abdominal obesity (waist circumference in men from Europe ≥ 94 cm, and in women ≥ 80 cm) and additionally co-existing two of the following abnormalities: triglycerides ≥ 150 mg/dl or dyslipidaemia related treatment cholesterol HDL < 40 mg/dl in males < 50 mg/dl in females or dyslipidaemia related treatment arterial pressure ≥ 130/85 mm Hg or arterial pressure related treatment fasting glycaemia ≥ 100 mg/dl or type 2 diabetes treatment
Assessment of metabolic syndrome | Second examination - at the end of the three-week program
  Metabolic syndrome (polymetabolic syndrome, syndrome X, insulin resistance syndrome, Reaven syndrome) - a set of interrelated factors significantly increasing the risk of atherosclerosis and type 2 diabetes, as well as their vascular complications.
  Abdominal (central) obesity
  At least three of the following five abnormalities must be identified to formulate a diagnosis:
  abdominal obesity (waist circumference in men from Europe ≥ 94 cm, and in women ≥ 80 cm) and additionally co-existing two of the following abnormalities: triglycerides ≥ 150 mg/dl or dyslipidaemia related treatment cholesterol HDL < 40 mg/dl in males < 50 mg/dl in females or dyslipidaemia related treatment arterial pressure ≥ 130/85 mm Hg or arterial pressure related treatment fasting glycaemia ≥ 100 mg/dl or type 2 diabetes treatment
Changes in blood parameter: TG | First examination - before the start of the rehabilitation program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  TG level:
  Below 150mg / dL (1.69mmol / L) Norm 150 - 199 mg / dL (1.69 - 2.25 mmol / L) Limit 200 - 499 mg / dL (2.26 - 5.63 mmol / L) High Above 500 mg / dL (5.64 mmol / L) Very high
Changes in blood parameter: TG | Second examination - at the end of the three-week program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  TG level:
  Below 150mg / dL (1.69mmol / L) Norm 150 - 199 mg / dL (1.69 - 2.25 mmol / L) Limit 200 - 499 mg / dL (2.26 - 5.63 mmol / L) High Above 500 mg / dL (5.64 mmol / L) Very high
Changes in blood parameter: atherogenic index | First examination - before the start of the rehabilitation program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  atherogenic index level
  * in men below 4.5 (below 3.5 after myocardial infarction)
  * in women below 4.0 (below 3.0 after myocardial infarction)
Changes in blood parameter: atherogenic index | Second examination - at the end of the three-week program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  atherogenic index level
  * in men below 4.5 (below 3.5 after myocardial infarction)
  * in women below 4.0 (below 3.0 after myocardial infarction)
Changes in blood parameter: CRP | First examination - before the start of the rehabilitation program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  CRP level:
  * CRP below 5 mg / l (up to 10 mg / l - in obese people with hypertension) norm
  * CRP above 40 mg / l - may indicate a mild viral infection or pregnancy;
  * CRP above 200 mg / l - bacterial inflammation develops in the body;
  * CRP above 500 mg / l - takes place in the situation of very serious infections with basic and bacterial infections and burns.
Changes in blood parameter: CRP | Second examination - at the end of the three-week program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  CRP level:
  * CRP below 5 mg / l (up to 10 mg / l - in obese people with hypertension) norm
  * CRP above 40 mg / l - may indicate a mild viral infection or pregnancy;
  * CRP above 200 mg / l - bacterial inflammation develops in the body;
  * CRP above 500 mg / l - takes place in the situation of very serious infections with basic and bacterial infections and burns.
Changes in blood parameter: serum glucose | First examination - before the start of the rehabilitation program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  serum glucose level: From 70 to 99 mg / dL (from 3.9 to 5.5 mmol / L) Normal glucose level From 100 to 125 mg / dL (from 5.6 to 6.9 mmol / L) Abnormal fasting glucose (pre-diabetes) From 126 mg / dL (7.0 mmol / L) Diabetes
Changes in blood parameter: serum glucose | Second examination - at the end of the three-week program
  Blood for the tests was drawn from basilic vein by medical personnel at the Rehabilitation Clinic.
  serum glucose level: From 70 to 99 mg / dL (from 3.9 to 5.5 mmol / L) Normal glucose level From 100 to 125 mg / dL (from 5.6 to 6.9 mmol / L) Abnormal fasting glucose (pre-diabetes) From 126 mg / dL (7.0 mmol / L) Diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Leszczak, PhD, Principal Investigator — Univeristy of Rzeszów,
Locations (1):
- University of Rzeszów, Rzeszów, Poland

REFERENCES:
- [Derived] Leszczak J, Pniak B, Gazda G, Guzik A. Assessment of the effects of rehabilitation of hand function using a biometrics device in people after stroke - a randomized controlled trial. Front Neurol. 2025 Sep 16;16:1643336. doi: 10.3389/fneur.2025.1643336. eCollection 2025. PMID 41036275